CLINICAL TRIAL: NCT04449497
Title: The 2020 Quality of Death and Dying Index
Acronym: QODDI
Status: Completed | Type: Observational
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Other Study IDs: S-20-110
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Palliative Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bereaved caregivers: Caregivers who, in the past two years,have lost a family member or close friend after a brief or extended period of illness or injury
- Country experts: Qualified individuals (providers, palliative care experts, policy makers) from countries across the globe with knowledge of the phenomenon of interest-end-of-life care.

SUMMARY:
Lien Centre for Palliative Care has been commissioned by Lien Foundation to produce the 2020 rankings of the Quality of End of Life Care across countries. This index will focus on patients with life limiting illnesses and their families and aims to produce an index and rankings that take into account the preferences of patients, their caregivers and providers in terms of what is truly important at end of life. The aim of this research is to investigate best practices in palliative care policy and implementation as they relate to end-of-life care for individuals with life-limiting or life-threatening conditions. This task will be completed through a systematic review of peer reviewed and grey literature, supplemented with qualitative interviews to identify the list of the candidate indicators to be used in the index. A final instrument when completed by country experts will allow for ranking countries in their ability to deliver high quality end of life care.

DETAILED DESCRIPTION:
Palliative care has gained considerable attention at the global, regional and national levels and there has been follow-up on actions outlined in the 2014 World Health Assembly (WHA) Resolution on palliative care. The WHA Resolution called countries to action to integrate palliative care into their national health strategies and as part of universal health coverage (UHC) efforts. Further, important contributions have been made to the literature on palliative care overall and at the end of life, such as by the Lancet Commission on Global Access to Palliative Care and Pain Relief as well as on quality healthcare.

Through this research, the Quality of Death and Dying Index will be published and it seeks to facilitate monitoring of country-level progress based on domains/sub-domains and indicators used to define quality of death and dying in the discourse on end-of-life care, and within the context of the contrasting realities occurring worldwide. Examining the various trajectories that countries have followed and the experiences of end-of-life care design and delivery by countries from different income groups and based on the viewpoint of diverse stakeholders will provide critical information for metrics development, namely the 2020 Quality of Death and Dying Index

ELIGIBILITY:
Inclusion Criteria for experts:

1. Technical expert with 10 or more years of experience in the field of palliative care and/or end-of-life care at the global, regional or national levels.
2. Current or former policy maker, at the state or national level and having actively engaged in development of policies and strategies on palliative care and/or end-of-life care.
3. Physicians, nurses and/or community health workers who have training to and have actively delivered end-of-life care.

For caregivers

1. In the past two years, lost a family member or close friend after a brief or extended period of illness or injury.
2. Involved in discussions with health care providers concerning the patient's choice of treatments
3. Involved in helping the patient receive medical care, such as accompanying the patient to doctor's visits.
4. Involved in looking after the patient's day to day well-being.

Exclusion Criteria:

* For patients 1. Individuals with physical, emotional or cognitive limitations which may prevent them from participating or comprehending the questions.

For all participants

1. Inability to understand English.
2. Minor and not below the age of 21 years.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will recruit caregivers of patients with life limiting illnesses as well as experts in the field of palliative care.
Sampling Method: Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Ranking of countries | 2 years
  Ranking of countries in their ability to deliver high quality end of life care.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No